CLINICAL TRIAL: NCT03557892
Title: Continuous Subcutaneous Insulin Infusion Associated With Continuous Glucose Monitoring in Comparison With Subcutaneous Multi-injection Insulin Therapy Using Degludec as Basal Insulin: a Randomized Crossover Trial in Type 1 Diabetes
Brief Title: Sensor-augmented Pump Versus Multiple Daily Injections With Degludec as Basal Insulin for Insulin Therapy in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Edoardo Mannucci, Director, Diabetology, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: T1DM001
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSII+CGM (Experimental)
  Interventions: Device: CGM+CSII
- MDI with degludec (Active Comparator)
  Interventions: Device: MDI with degludec

INTERVENTIONS:
Device: CGM+CSII — Animas Vibe Platinum insulin pump and Dexcom G4 CGM
  Arms: CSII+CGM
Device: MDI with degludec — Multiple injection therapy with any short-acting analogue as bolus insulin and degludec as basal insulin
  Arms: MDI with degludec

SUMMARY:
Several studies have shown that Continuous Subcutaneous Insulin Infusion together with Continuous Glucose Monitoring improves glycemic control in type 1 diabetes when compared to more traditional approaches; however, in available trials the basal insulin used in multi-injection therapy is typically glargine, which is associated with a higher hypoglycemic risk than degludec.

This study will assess the efficacy and safety of Continuous Subcutaneous Insulin infusion (CSII) combined with Continuous Glucose Monitoring (CGM), as compared to Multiple Daily Injections (MDI) of insulin analogues, using degludec as basal insulin, associated with traditional self-monitoring of capillary blood glucose (SMBG) in patients with type 1 diabetes. A crossover design was chosen in order to minimize study sample improving statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Duration of diabetes > 2 years
* Current treatment with MDI, using insulin analogues as bolus and basal insulin
* HbA1c<64 mmol/mol

Exclusion Criteria:

* HbA1c>64 mmol/mol
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetologia AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Subcutaneous Insulin Infusion+Continuous Glucose Monitoring (CSII+CGM): CGM+CSII: Animas Vibe Platinum insulin pump and Dexcom G4 CGM
- Multiple Daily Injections Regimen (MDI) With Degludec: MDI with degludec: Multiple injection therapy with any short-acting analogue as bolus insulin and degludec as basal insulin
Period: Overall Study
Arm/Group | Continuous Subcutaneous Insulin Infusion+Continuous Glucose Monitoring (CSII+CGM) | Multiple Daily Injections Regimen (MDI) With Degludec
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSII+CGM | MDI With Degludec | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [22 to 71] | 41 [21 to 72] | 42 [21 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 61 (4) | 62 (5) | 61 (5)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Variation of HbA1c in each treatment phase (difference between end-of-treatment and baseline for each treatment phase)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | CSII+CGM | MDI With Degludec
Number analyzed (Participants) | 14 | 14
mmol/mol | -6.1 (4.0) | 0.5 (4.5)

2. Secondary Outcome: Severe Hypoglycemia
Description: Number of subjects with at least one episode of severe hypoglycemia, for each treatment phase
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | CSII+CGM | MDI With Degludec
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

3. Secondary Outcome: Local Reactions
Description: Number of participants with local reactions at infusion/glucose monitoring site
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | CSII+CGM | MDI With Degludec
Number analyzed (Participants) | 14 | 14
Participants | 8 | 0

ADVERSE EVENTS:
Time Frame: 4 months for each treatment arm
Arm/Group | CSII+CGM | MDI With Degludec
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 8/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSII+CGM (N=14) | MDI With Degludec (N=14)
Local skin reactions (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03557892/Prot_SAP_000.pdf